CLINICAL TRIAL: NCT05497219
Title: Establishing Reference Values and Clinical Decision Points for Quantitative Videofluoroscopic Measures of Swallowing
Brief Title: Reference Values for Videofluoroscopic Measures of Swallowing
Acronym: NIA_RV
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Florida (Other); McMaster University (Other); National Institute on Aging (NIA) (NIH); Ohio State University (Other); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 21-6019; R01AG077481 (NIH)
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Dysphagia, Oropharyngeal
Keywords: Deglutition
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy adults (Other): Adults aged 18 or older with no history of swallowing impairment
  Interventions: Diagnostic Test: Videofluoroscopic Swallowing Study (VF)
- Parkinson Disease (Other): Adults with a neurologist-confirmed diagnosis of Parkinson Disease who also report symptoms of swallowing impairment, defined as a score >/= 200 on the Sydney Swallow Questionnaire.
  Interventions: Diagnostic Test: Videofluoroscopic Swallowing Study (VF)
- Chronic Obstructive Pulmonary Disease (Other): Adults with a respirologist-confirmed diagnosis of Chronic Obstructive Pulmonary Disease who also report symptoms of swallowing impairment, defined as a score >/= 200 on the Sydney Swallow Questionnaire.
  Interventions: Diagnostic Test: Videofluoroscopic Swallowing Study (VF)
- Acute Stroke (Other): Adult inpatients in the acute stage post stroke who are referred for swallowing assessment.
  Interventions: Diagnostic Test: Videofluoroscopic Swallowing Study (VF)

INTERVENTIONS:
Diagnostic Test: Videofluoroscopic Swallowing Study (VF) — A videofluoroscopy (VF) is a dynamic radiological evaluation of swallowing in which the participant swallows liquid or food boluses of different consistencies prepared with barium contrast. The x-rays are recorded at 30 frames per second.

SUMMARY:
Dysphagia (swallowing impairment) is a serious health condition seen in many age-related disease and injury processes. Although videofluoroscopy (VF) is an international "gold standard" dysphagia diagnostic exam, there is a paucity of available normative physiologic VF reference values in healthy adults across the age span to guide interpretation of these examinations. In this project, the investigators will extend previous work on the quantitative measurement of swallowing physiology from VF examinations to establish reference values for swallowing in healthy adults, and to identify clinical decision point values for differentiating healthy swallowing across the age span from disordered swallowing in several high-risk clinical populations to study dysphagia.

DETAILED DESCRIPTION:
Dysphagia (swallowing impairment) is a serious health condition seen in many age-related disease and injury processes. Although videofluoroscopy (VF) is an international "gold standard" dysphagia diagnostic exam, there is a paucity of available normative physiologic VF reference values in healthy adults across the age span to guide interpretation of this examination. This fundamental gap in knowledge contributes to poor agreement in the identification of swallowing impairment and its underlying mechanisms. To enable better dysphagia diagnostics, there is a critical need to establish reference values for VF swallowing measures across the healthy age span.

In a previous study, the investigators developed a rigorous method for measuring swallowing physiology from VF: the Analysis of Swallowing Physiology: Events, Kinematics and Timing (ASPEKT Method). That study led to publication of initial ASPEKT reference values from 40 young healthy adults (<60 years) and preliminary analyses comparing data from healthy older adults and small cohorts of adults with dysphagia to these reference data.

In this project, the investigtors will:

* validate the ASPEKT Method healthy reference values for swallowing across the adult life span; and
* profile swallowing patho-physiology in clinical groups where dysphagia is a cause of morbidity to identify clinical decision points that can be used for diagnosis and outcome measurement.

This study will explore the following research questions:

Research Question 1: Will > 5% of healthy adult participants in a new sample show ASPEKT values outside the common reference interval calculated in a prior sample? • VF measures will be collected in a prospective sample of 280 healthy adults, controlling for sex, age, and bolus consistency. Updated reference interval boundaries for healthy swallowing will be calculated.

Research Question 2: Do specific clinical conditions present with specific patterns of swallowing pathophysiology?

• VF measures will be prospectively collected in 3 high-risk dysphagia cohorts: adults with Parkinson Disease, Chronic Obstructive Pulmonary Disease, adults in the acute stage post-stroke. Values for these clinical cohorts will be compared to age- and sex-matched reference values from healthy participants. This will delineate swallowing impairment profiles to inform clinical decision points for diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Volunteers: no history of swallowing difficulties.
2. Clinical cohorts: physician confirmed diagnosis of the condition of interest plus symptoms of swallowing difficult, defined as a score >/=200 on the Sydney Swallow Questionnaire.

Exclusion Criteria:

* cognitive communication difficulties that may hinder comprehension of the study documents
* known allergies to latex, due to the possibility that these items will come into contact with the oral mucosa during data collection
* current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with unsafe swallowing | Baseline
  Swallowing safety requires the ability to protect the airway to prevent penetration-aspiration (the entry of food or liquid material into the airway during swallowing). Swallowing safety will be measured using the Penetration-Aspiration Scale, an 8-point categorical scale which captures the depth to which any material enters the airway and whether or not the material is ejected. Levels 1 and 2 on the scale are considered safe, while levels > 2 are considered unsafe. Actual scale scores (1-8) will be recorded and then converted to binary categorical scores (< 3 vs >/= 3). The frequency (count) of participants showing scores > 2 will be reported by bolus consistency (thin, slightly thick, mildly thick, moderately thick and extremely thick liquids).
Number of participants with impaired swallowing efficiency | Baseline
  Swallowing efficiency requires the ability to move a bolus of food or liquid from the mouth through the pharynx into the esophagus in a single swallow without leaving residue behind in the pharynx. Residue is material remaining behind in the pharynx after the swallow. Residue will be measured by tracing the area of barium visible on a lateral view x-ray (in pixels, using ImageJ software) and dividing that area by the squared length of the C2-C4 cervical spine. This cervical spine scalar provides a common anatomical reference that is a proxy for pharyngeal size, and enables the comparison of residue severity across different people with different neck length and pharynx size. In healthy swallowing, residue is expected to be minimal, i.e. less than 1% (C2-4)squared. The frequency (count) of participants showing residue above this threshold will be reported by bolus consistency (thin, slightly thick, mildly thick, moderately thick and extremely thick liquids).
Number of participants with delayed airway closure ("Time-to-laryngeal-vestibule-closure") | Baseline
  Swallowing safety requires the ability to protect the airway to prevent penetration-aspiration (the entry of food or liquid material into the airway during swallowing). Closure of the entrance to the airway ("laryngeal vestibule closure" or LVC) must be achieved in a timely manner. Time-to-LVC will be measured, i.e., the time interval between onset of the pharyngeal swallow (i.e. onset of the hyoid burst movement) and the first frame showing the most-complete closure of the laryngeal vestibule. In healthy adults, the upper limits (97.5th percentile value) for this measure are currently reported to be 267 ms on thin liquids, 367 ms on slightly thick liquids, 367 ms on mildly thick liquids, 300 ms on moderately thick liquids and 267 ms on extremely thick liquids. The frequency (count) of participants displaying time-to-LVC measures above these limits will be reported by bolus consistency (thin, slightly thick, mildly thick, moderately thick and extremely thick liquid).
Number of participants with poor pharyngeal constriction | Baseline
  Efficient clearance of a bolus of food or liquid through the pharynx in swallowing requires constriction of the pharynx. In healthy adults, there is typically no unobliterated space visible in the pharynx on a lateral view x-ray image on the frame of maximum constriction. ImageJ software will be used to measure the area of unobliterated pharyngeal space, which is expressed as a % of an anatomical reference scalar defined as the squared length of the C2-C4 cervical spine [%(C2-4)squared]. Larger unobliterated area reflects impairment in pharyngeal constriction. In healthy adults, the upper limits (97.5th percentile) for this measure are currently reported to be 6.2%(C2-4)squared on thin, 5% on slightly thick, 7.5% on mildly thick, 4.9% on moderately thick and 3.8% on extremely thick liquids. The frequency (count) of participants with pharyngeal constriction area above these limits will be reported by bolus consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Catriona M Steele, PhD, Principal Investigator — University Health Network, Toronto; Emily K Plowman, PhD, Principal Investigator — Ohio State University
Locations (5):
- United States (3):
  - University of Florida, Gainesville, Florida
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
- Canada (2):
  - McMaster University, Hamilton, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No